CLINICAL TRIAL: NCT03349827
Title: A Study of Conversion Therapy Using Hyperthermic Intraperitoneal Chemoperfusion (HIPEC) and Systemic Oxaliplatin/S1 Chemotherapy Combined With Apatinib in Unresectable Peritoneal Metastases From Gastric Cancer
Brief Title: HIPEC and Systemic Chemotherapy Combined With Apatinib in Unresectable Peritoneal Metastases From Gastric Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrolled patients received the second surgery.
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Bin Xiong, MD, Zhongnan Hospital, Wuhan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WuhanU_Peritoneal Metastases
Record Dates: First submitted 2017-11-09; First posted 2017-11-22 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Peritoneal Metastases From Gastric Cancer
MeSH Terms: interventions — Laparotomy; Hyperthermic Intraperitoneal Chemotherapy; Neoadjuvant Therapy; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): HIPEC with Docetaxel/ Lobaplatin at the time of fist surgery and twice repeat within one week after the surgery, following 2 cycles of 3-week Oxaliplatin/S1 chemotherapy combined with Apatinib and 1 cycles of 3-week Oxaliplatin/S1 chemotherapy. The second surgery, exploratory laparoscopy or laparotomy, is carried out one week later after the series of systemic chemotherapy.
  Interventions: Procedure: exploratory laparoscopy or laparotomy; Procedure: HIPEC; Drug: Systemic chemotherapy; Drug: Apatinib

INTERVENTIONS:
Procedure: exploratory laparoscopy or laparotomy — Exploratory laparoscopy or laparotomy, for PCI score or radical gastrectomy and cytoreductive surgery
Procedure: HIPEC — Normal saline 3000ml-4000ml, Docetaxel 50mg/m2, Lobaplatin 50mg/m2, 43°C, 60min.
Drug: Systemic chemotherapy — Oxaliplatin: 130mg/m2, day 1. S1: 60mg, twice daily, day 1 to day 14. S1:60mg twice daily for two weeks, and then suspend for one week
  Other Names: SOX
Drug: Apatinib — 500mg, once daily, day 1 to day 21.

SUMMARY:
The prognosis of patients with unresectable peritoneal metastases from gastric cancer is poor. These patients may obtain survival benefit from radical gastrectomy and cytoreductive surgery (CRS). The response rates of previous conversion therapy are low. Hyperthermic intraperitoneal chemoperfusion (HIPEC) and systemic chemotherapy are effective methods of reducing peritoneal cancer index (PCI) levels. Apatinib, a novel targeted inhibitor of VEGF receptor 2 (VEGFR2), shows significant antitumor activity in the patients with gastric cancer. The purpose of this study is to investigate the efficacy and safety of HIPEC and systemic chemotherapy combined with Apatinib in the conversion therapy of peritoneal metastases from gastric cancer.

DETAILED DESCRIPTION:
To determine the efficacy and safety of HIPEC and systemic chemotherapy combined with Apatinib in the conversion therapy of peritoneal metastases from gastric cancer, patients undergo HIPEC with Docetaxel/ Lobaplatin at the time of fist surgery and twice repeat within one week after the surgery, following 2 cycles of 3-week Oxaliplatin/S1 chemotherapy combined with Apatinib and 1 cycles of 3-week Oxaliplatin/S1 chemotherapy. The second surgery, exploratory laparoscopy or laparotomy, is carried out one week later after the series of systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological proved diagnosis of gastric cancer.
* Unresectable peritoneal metastases and primary tumor proved at surgery.
* No evidence of distant metastases.
* Have not received radiotherapy, chemotherapy or immunotherapy.
* ECOG score: 0~2.
* Written informed consent is obtained prior to commencement of trial treatment.

Exclusion Criteria:

* Existence of distant metastasis outside the abdomen.
* Any previous radiotherapy, chemotherapy or immunotherapy.
* Active systemic infections.
* Inadequate cardiac function, renal function, liver function or bone marrow function at the beginning of the trial.
* Female patients who are pregnant or breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
radical resection rate | 3 months
  The rate between the number of patients with radically resectable peritoneal metastases and those with unresectable peritoneal metastases

SECONDARY OUTCOMES:
the Peritoneal Cancer Index score | 3 months
  The score range from 0 to 39, higher values represent a worse outcome
overall survival | 3 years
  The overall survival time
complication rate | 3 years
  The rate of adverse complication

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan University, Wuhan, Hubei, China